CLINICAL TRIAL: NCT03588364
Title: The Role of Osteopathic Manipulation in the the Management of Post-traumatic Migraine
Acronym: OMT/mTBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Hollis King, Health Sciences Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: OMT/mTBI
Record Dates: First submitted 2018-07-04; First posted 2018-07-17 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Migraine Disorders; Post-Traumatic Headache
Keywords: osteopathic manipulation
MeSH Terms: conditions — Migraine Disorders; Post-Traumatic Headache | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: This is a 30-week prospective, randomized delayed treatment control group design in which 20 participants from the community will be randomized 1:1 into (a) an immediate treatment group that will receive 12 weeks of osteopathic manipulation (OMT) treatment plus standard of care right away or (b) delayed treatment group that will receive 12 weeks of OMT plus standard of care after a 6-week waiting period. The delayed treatment group initially serves as a control condition but then receives the experimental treatment.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the study coordinator and the participants are privy to the assigned treatment arm (immediate vs. delayed) until the study is complete and the database is locked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathic Manipulation (Experimental): Twelve weekly sessions using the techniques of osteopathy in the cranial field.
  Interventions: Other: Osteopathic Manipulation
- Waitlist Control (No Intervention): Six-week waiting period.

INTERVENTIONS:
Other: Osteopathic Manipulation — Osteopathic manipulation involves a number of different manual techniques. These include muscle inhibition; myofascial release; muscle energy stretch; counterstrain; facilitated positional release ; osteopathy in the cranial field ; balanced ligamentous tension/ligamentous articular strain; one or all of these techniques may be used. Participants will be positioned on an exam table supine, seated, lateral decubitus, prone, or in their position of greatest comfort for the procedure.
  Arms: Osteopathic Manipulation

SUMMARY:
This study evaluates the use of osteopathic manipulation (manual medicine) for migraine headache following traumatic head injury. Headache is an important and very common somatic complaint among people with traumatic brain injury and an important cause of disability in the United States. Over 15-percent of soldiers deployed to Iraq sustained concussion. A majority of these patients suffer from headaches. Many of these are classified as migraine headache that do not respond to medications. Osteopathic manipulation is practiced by physicians in the United States and has been shown to be beneficial in some migraine patients. However, its use in the management of persistent post-traumatic headaches has not been explored. The investigators will use a randomized cross-over design to evaluate post-traumatic migraine patients' response to osteopathic manipulation.

DETAILED DESCRIPTION:
This is a 30-week prospective, randomized delayed treatment control group design in which 20 participants from the community will be randomized 1:1 into (a) an immediate treatment group that will receive 12 weeks of osteopathic manipulation (OMT) treatment plus standard of care right away or (b) delayed treatment group that will receive 12 weeks of OMT plus standard of care after a 6-week waiting period. The delayed treatment group initially serves as a control condition but then receives the experimental treatment. The investigators selected this control condition to improve our statistical power in this small pilot study. As noted, all participants will continue to receive standard of care throughout the study as a washout is not feasible with osteopathic manipulation and removing standard of care could exacerbate the participant's symptoms. Participants in both arms will be followed for another 12 weeks after the 12 weeks of OMT, resulting in 24 weeks of study participation for the immediate treatment group and 30 weeks of study participation for the delayed treatment group, with participants in both arms answering a series of questionnaires to evaluate migraine frequency and impact, treatment efficacy, side effects, adherence t standard of care and depressive symptoms every 6 weeks throughout their study participation. Participant encounters will consist of screening, psychometric and functional scale administration at every 6 weeks for a total of 24-30 weeks, as well as 12 weeks of OMT treatments for participants in both study arms. Study participants will likely come from UCSD internal referrals.

ELIGIBILITY:
Inclusion Criteria:

* History of TBI, concussion, post-concussive syndrome
* Headache frequency >/equal 4 per month
* Post-traumatic headache, migraine type
* MIDAS Grade I-IV
* Headaches continue to occur 3 months to 1 year after the injury
* No history of uncontrolled migraine prior to head injury

Exclusion Criteria:

* Headache medication change (Tricyclic antidepressant, antiepileptic medication, propranolol, verapamil, duloxetine, butterbur, Botox) within 30 days
* Non-pharmacologic headache management change (reduction in caffeine intake, reduction in alcohol intake, sleep hygiene, exercise) within 30 days
* Less than 3 months from injury
* History of uncontrolled migraine prior to TBI
* Currently taking oral anti-coagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Headache Frequency Log | 6 weeks
  Participants will complete a form indicating the frequency, location, duration, characteristics, and associated features of their headache.

SECONDARY OUTCOMES:
Migraine Disability Assessment Score (MIDAS) | 6 weeks
  Scale measures migraine disability by asking participants to indicate number of various events missed (or completed with reduced productivity) over the past three months; as well as average pain associated with headaches in the past 3 months.
Center for Epidemiological Studies-Depression (CES-D) | 6 weeks
  20-item measure that asks respondents to rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
36-Item Short Form Survey Instrument (MOS-SF-36) | 6 weeks
  36-item, patient-reported survey of health-related quality of life. Each of the eight scales is transformed into a 0-100 scale. The 8 scales include: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Hollis H King, DO, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No